CLINICAL TRIAL: NCT02860975
Title: Physiological and Biochemical Response to Prolonged Exposure to Hypoxic Breathing in Healthy Volunteers
Brief Title: Prolonged Hypoxic Breathing in Healthy Volunteers: a Safety Study
Acronym: MGH-nitrogen
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data analysis completed after half volunteers were enrolled
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Rezoagli, Emanuele, M.D., Massachusetts General Hospital, Harvard Medical School (Unknown); Ferrari, Michele, M.D., Massachusetts General Hospital, Harvard Medical School (Unknown); Patel, Sarvagna, B.A., Massachusetts General Hospital, Harvard Medical School (Unknown); Zapol, Warren M., M.D., Massachusetts General Hospital, Harvard Medical School (Unknown); Fisher, Daniel, R.R.T., Massachusetts General Hospital, Harvard Medical School (Unknown); Jain, Isha, B.A., Massachusetts General Hospital, Harvard Medical School (Unknown); Mootha, Vamsi, M.D., Massachusetts General Hospital, Harvard Medical School (Unknown); Harris, Stuart N., M.D., Massachusetts General Hospital, Harvard Medical School (Unknown); Karaa, Amel, M.D., Massachusetts General Hospital, Harvard Medical School (Unknown)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Assistant Professor of Anesthesia, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGH-ACCCR
Record Dates: First submitted 2016-07-30; First posted 2016-08-10 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Prolonged Hypoxia; Safety; Mitochondrial function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhaled Nitrogen (Experimental): A humidified mixture of gas will be delivered by mask, nasal cannulae, and small room-sized tent. Inspiratory oxygen fraction (FiO2) will be gradually decreased to 11% over a period or five days to obtain a peripheral capillary O2 saturation (SpO2) between 80%-85% (corresponding to 40-55 mmHg of arterial partial oxygen pressure (PaO2)). Healthy volunteers will be monitored and blood and urine will be obtained at 24h and 48 hours after returning to normoxia.
  Interventions: Other: Inhaled Nitrogen

INTERVENTIONS:
Other: Inhaled Nitrogen — To create the correct gas mixture, nitrogen tanks or membrane technology nitrogen generators will be utilized.
  Humidified, high flow, hypoxic gas by nasal cannula will allow the participant to walk short distances, eat, execute basic personal needs (e.g., use of toilette, washing, bathing etc.), or take breaks from wearing the mask.

SUMMARY:
The purpose of this study is to define the safety and the biochemical-physiological response of prolonged exposure to a normobaric low-oxygen environment in healthy volunteers.

DETAILED DESCRIPTION:
The primary endpoint of this research study is to prove safety in healthy subjects breathing humidified hypoxic inspiratory gas mixture for 5 days.

The secondary endpoint of our study is to describe the physiological and biochemical changes during the 5-day hypoxic period and the 2 days after return to normoxia.

The specific aims are as follows:

AIM 1: To provide a safe, controlled setting for prolonged exposure of monitored healthy adults to a normobaric, low-oxygen environment for five days.

AIM 2: To carry out a seven-days long pilot safety-study in twelve healthy young subjects by inducing hypoxia with a humidified normobaric gas mixture containing oxygen (O2) content as low as 11% to reach a peripheral oxygen saturation (SpO2) between 80%-85%.

Screening will consist of a physical examination, 12-lead electrocardiogram, cardiac echocardiography, sickle cell screening test, and current (within 12 weeks of clearance exam with no intervening medical treatment) routine blood and urine analyses.

Women using oral, subdermal or injectable contraceptives, and those using other means of birth control may participate. A urine pregnancy test will be conducted as part of the screening process for study participation no more than 7 days before starting the study and it will be repeated on the day of enrollment. The test result will be read by a female staff member who will keep the result confidential. If a woman declines to have a pregnancy test, she will not be able to participate.

Recruitment will be done in three ways:

1. Broadcast MGH: Research Studies In Need of Volunteers
2. Enrollment in the Research Study Volunteer Program (RSVP) for Health of Massachusetts General Hospital (MGH) and Brigham Women Hospital (BWH)
3. Advertising at the Partners clinical trials Potential study subjects will be able to contact study investigators by phone or email to verify eligibility according to the inclusion/exclusion criteria and to set up the first visit, at which point the study will be explained in detail and they will be asked to provide informed consent. Subjects may contact the study investigators at any time to withdraw from the study. Confidentiality will be preserved to the fullest extent.

The study will be explained to each volunteer in detail. Signing of an Informed Consent Form will be requested for participation in the study. Volunteers will sign the informed consent at the beginning of the study. The Principal Investigator (PI) and/or Co-PIs of the study will be available to answer any questions the volunteer may have. Consent can be withdrawn at any time. The investigators will access personal Medical Information (PMI) for study purposes. There is no randomization in this interventional physiological study. All patients will receive the same procedures in the same order.

Biostatistical analysis:

A de-identified code will be assigned to the patient and registered on a dedicated enrollment log. The baseline study volunteer data (vital signs and biochemical measurements) will be collected from the MGH electronic medical chart (EPIC). Prospective collection of patient data will include specific data sheet. Data will be expressed as means ± standard deviation (SD) or median/interquartile range (IQR) as appropriate.

Sample size: this research-project is aimed to study 12 healthy subjects for the entire 7-day study period. To account for possible dropouts and missing data, up to 18 healthy volunteers will be enrolled.

Sample size calculation: This is an intra-hospital safety trial with the purpose of testing methods to re-create a safe hypoxic environment for possible future studies in patients with mitochondrial dysfunction. While 2 or 3 subjects would likely be sufficient to test our methods to reliably delivery humidified nitrogen (N2) and (O2) in predetermined concentrations, this method will be tested in 12 healthy subjects to reproduce our methods and obtain feedback from the volunteers. To account for possible dropouts, up to 18 healthy volunteers will be enrolled.

Risk and discomforts

1. Complications of surgical and non-surgical procedures, etc. Participants in the study will undergo 3 procedures during the study: hypoxic gas administration, phlebotomy, and echocardiography.

   * Facemask.

     1. Claustrophobia is one of the exclusion criteria. If a subject develops claustrophobia, he/she may leave the trial at any point.
     2. The most common side effects of facemask are pressure related, such as redness, irritation over the mask's borders. To decrease possible skin irritation and abrasions, subjects will be using a tent during the night and high flow nasal cannula during the day for breakfast, lunch and dinner. Additionally they will be able to choose whether to use high-flow nasal cannula or the facemask during the day at any time as an alternative to the facemask.
   * Tent. Risks associated with use of tents include unintended hypoxia, hypercarbia, and claustrophobia. These tents are made at the MGH shop and routinely used on the burn unit to maintain elevated temperature (80-90 °F) and humidification in critically ill patients. Our subjects will be continuously monitored for hypoxia and clinical condition to limit risk of unintended hypoxia or hypercarbia. Claustrophobia will be handled as described previously.
   * Nasal cannula and non-invasive high flow humidified gas. All participants will wear non-invasive high flow humidified gas for part of study period. Unlike masks, high flow nasal cannula is well tolerated in hospitalized patients and warm humidified air alleviates discomfort of the high flow. In order to avoid abrasions, we will inspect subjects' nasal mucosa in the morning and evening.
   * Intravenous (IV) punctures and phlebotomy. Risks related to phlebotomy include bruising, hematoma formation, cellulitis, superficial thrombosis, bleeding and phlebitis. An IV nurse or an anesthesiologist will perform phlebotomy to minimize subject discomfort.
   * Trans-thoracic echocardiography. Echocardiography will be performed on daily basis: Echocardiographic assessment of pulmonary artery pressure and cardiac output is a noninvasive and painless maneuver. It is commonly used in clinical practice, has been used in the field under hypoxic conditions, and is safe for the study subjects. If the echocardiographic study reveals any unexpected cardiac disease the subjects will be informed and also their primary care physician (PCP) will be informed. If the subject does not have a PCP, we will provide information about choosing a PCP.

   In presence of an abnormal physical exam and/or additional abnormal laboratory results (including a positive pregnancy test), subjects will be informed.
2. Drug side effects and toxicities

   A gas mixture enriched with nitrogen will be tested. It is expected that subjects may suffer to a certain degree of acute mountain sickness. Symptoms may include: headache, dizziness, poor sleep, poor appetite and fatigue that are related to hypoxia. These symptoms are well described in mountain climbers and will not require interruption of the study, unless the subject requests exiting the study. Furthermore, in this proposed model of normobaric hypoxia, the risk of acute mountain sickness symptoms has been reported to be lower than hypobaric hypoxia (simulated altitude). The following risks might also occur:
   * Risks Associated with Hypoxia: Severe hypoxemia (SpO2 ≤ 70%), especially with decreased respiratory rate can ensue. Since the fraction of inspired of oxygen can be quickly increased, there is no risk of developing prolonged hypoxia events. If SpO2 ≤ 70% decreases for more than one continuous minute, nitrogen administration will be stopped and the fraction of inspired of oxygen will be increased to 50%. The study will be stopped. Symptoms of hypoxia (light headedness, dizziness) typically resolve immediately upon return to a normal range of SpO2. If hypoxia symptoms are present, subjects will exit the study only after all symptoms of light-headedness or dizziness are resolved, and headache or nausea is absent.
   * Acute mountain sickness can very rarely progress to high altitude pulmonary edema (HAPE) or high altitude cerebral edema (HACE) and would be case reportable were either to occur in normobaria at the limited hypoxic challenge we will be employing. Though HAPE is very unlikely to occur, we will provide daily monitoring by echocardiography, clinical exam (auscultation for rales and unusual dyspnea at rest solicited), and pulse oximetry. If HAPE does occur, the study will stop and the subject treated with oxygen until resolution of symptoms.
   * HACE is also a very unlikely potential risk in this study. If a subject develops any evidence of ataxia or altered mental status, they will be immediately withdrawn from the study. FiO2 will be increased to 50%, dexamethasone 8 mg IV will be administered, and head computed tomography (CT) will be performed to rule out other much more common sources (e.g. spontaneous subarachnoid hemorrhage) of these complaints. If no CT abnormalities are noted, a brain magnetic resonance imaging (MRI) will be obtained to assess for cerebral edema and characteristic T2 weighted signal change in the corpus callosum consistent with HAPE..

   Any study subject who experiences side effects sufficient to prompt premature termination of the study will not be allowed to continue in the protocol. He or she will be monitored until vital signs normalize and transthoracic echocardiography (TTE) shows normal right heart function.
3. Device complications/malfunctions Nitrogen generator: If the nitrogen generator is malfunctioning, air will be enriched with nitrogen from nitrogen-tanks. The manufacturer will be contacted (Higher Peak LLC, Winchester, Massachusetts (MA) 01890) in order to deliver a new nitrogen generator.
4. Psychosocial (non-medical) risks Psychosocial risks include prolonged indoor exposure and perceived isolation from a subject's daily routine, family and friends. Subjects will have ready access to their personal communication devices (e.g. smart phone for voice/ social media use) during times when they are not actively participating in testing procedures. Subjects may be visited in person on the study floor. We do not anticipate any other psychosocial risks to the study subjects from participation in this protocol. Strict confidentiality will be maintained by the research team at all times, including keeping all data in a secure, locked cabinet with limited access. All specimens will be coded after they are obtained and the code key kept in a locked cabinet. All electronic data will be stored in a Partners encrypted laptop. Samples given to parties outside of MGH for analysis will be coded to maintain confidentiality.

Monitoring and Quality Insurance:

Due to the small size of the study, no independent monitoring is deemed necessary. The PI himself will be responsible for the monitoring of the study.

The PI and co-Is will be responsible for the monitoring of the study. Dr. Lorenzo Berra is the Principal Investigator and he is an Anesthesiologist and Intensivist at MGH and Assistant Professor at Harvard Medical School.

Stopping rules

The principal investigator and co-investigators will perform the review and decision regarding altering or stopping the protocol. Mild or moderate adverse events will be presented in progress reports at continuing reviews. Protocol exit criteria will be:

* Desaturation: SpO2<70% for more than 1 minute not immediately responsive to oxygen therapy.
* Chest pain with evidence of ischemia on electrocardiography (EKG) (e.g., T-wave inversions, ST segment changes).
* Signs and symptoms of acute pulmonary edema:

  * Rapidly progressive, severe shortness of breath at rest..
  * Severe dyspnea, or a feeling of suffocating or drowning despite return to normoxia.
  * Wheezing or gasping accompanied with anxiety, restlessness or a sense of apprehension.
  * A cough that produces frothy sputum that may be tinged with blood
* Signs and symptoms of acute cerebral edema:

  * acute ataxia or altered mental status
  * any focal neurologic deficit.
* Increase in systolic pulmonary artery pressure of 15 mmHg from baseline (first trans-echocardiography in ambient air)
* Syncope.
* Febrile illness (> 100.4 on two contiguous assays 1 hour apart)
* Subject may voluntarily withdraw from the study at any time.

ELIGIBILITY:
Inclusion criteria

* Have a photo identification (ID)
* Male or female individuals age between 18 and 40 years old
* BMI between 19 and 24.9 kg/m2
* Having capacity to consent to the study Exclusion criteria
* Evidence of any physical, mental, and/or medical conditions that would make the proposed studies relatively more hazardous
* Prior high altitude pulmonary edema (HAPE) or high-altitude cerebral edema (HACE) diagnosis
* Born at altitudes greater than 2,100 m (~7,000 ft)
* Systemic disease with or without any functional limitation; including

  * controlled hypertension
  * controlled diabetes without systemic effects
* Pregnancy determined by urine pregnancy test, detecting presence of human chorionic gonadotropin (hCG), or less than six weeks postpartum
* Women who are not willing to receive urine pregnancy tests
* Active smoking. Volunteers may be enrolled if they quit smoking for more than 1 year.
* Excess alcohol use: more than ½ L/day of wine consumption or equivalent
* Any current medication use except oral contraceptives.
* Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas that are more than 1,200 m for more than four days within the last 2 months
* Tobacco chewers
* Abnormal hemoglobin or hematocrit levels or presence of hemoglobin S
* Evidence of apnea or other sleeping disorders
* Evidence of asthma
* Lower respiratory infection within the last 30 days
* If applicable, unwilling to refrain from using energy drinks or other caffeinated beverages for 7 days prior to and during the study
* If applicable, unwilling to refrain from use of all over-the-counter oral medications, herbal remedies, and nutritional supplements for 7 days prior to and during the study
* Not willing to have blood drawn from an arm vein each test day of the study
* Claustrophobia (inability to wear a facemask) or other active psychiatric conditions or not willingness to cooperate with the investigators and the other medical team
* Currently enrolled in another research study
* Facial abnormalities that would preclude proper use of a face mask

Pregnancy Prevention/Testing: Women using oral, subdermal or injectable contraceptives, and those using other means of birth control may participate. A urine pregnancy test will be conducted as part of the screening process for study participation no more than 7 days before starting the study. The test result will be read by a female staff member who will keep the result confidential. If a woman declines to have a pregnancy test, she will not be able to participate.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Peripheral oxygen saturation | 7 days
  Peripheral oxygen saturation of the healthy volunteers receiving different levels of FiO2 will be continuously monitored for the 5 days of hypoxia titration and the 2 days after return to normoxia.

SECONDARY OUTCOMES:
Erythropoiesis | 7 days
  Erythropoietin will be tested each day during the 7 day study period.
Pulmonary pressure | 7 days
  Pulmonary pressure will be non-invasively measured via transthoracic echocardiography each day during the 7 day study period.
Mitochondrial oxidative stress | 7 days
  Plasma reactive oxygen species (ROS) will be evaluated each day during the 7 day study period.
Acid-base status | 7 days
  Venous acid-base status will be evaluated each day during the 7 day study period.
Systemic blood pressure | 7 days
  Systemic blood pressure will be regularly monitored during the 7 day study period.
Heart rate | 7 days
  Heart rate will be continuously monitored via electrocardiography (EKG) during the 7 day study period.
Respiratory rate | 7 days
  Respiratory rate will be regularly monitored during the 7 day study period.
Anaerobiotic glycolytic pathway | 7 days
  Lactate levels will be tested each day during the 7 day study period.
Energy metabolism | 7 days
  Alpha-hydroxybutyrate levels will be tested each day during the 7 day study period.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Inhaled nitric oxide selectively reverses human hypoxic pulmonary vasoconstriction without causing systemic vasodilation. — http://www-ncbi-nlm-nih-gov.ezp-prod1.hul.harvard.edu/pubmed/8457043
- See also: Hypoxia as a therapy for mitochondrial disease. — http://www-ncbi-nlm-nih-gov.ezp-prod1.hul.harvard.edu/pubmed/26917594
- See also: Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. — http://www-ncbi-nlm-nih-gov.ezp-prod1.hul.harvard.edu/pubmed/24285617